CLINICAL TRIAL: NCT05239377
Title: Clinical Evaluation of the Benefits of the MiProstate Platform: Follow-up Study
Brief Title: MiProstate - Information Hub for the Prostate Cancer Care Flow
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Principal Investigator, Olof Akre, Professor, Karolinska University Hospital
Other Study IDs: MiProstate
Record Dates: First submitted 2022-01-10; First posted 2022-02-14 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Baseline: Pre-prostatectomy conferences conducted without the use of digital support
- ISPM -MiProstate: Pre-prostatectomy conferences conducted with the use of digital support (ISPM- MiProstate)
  Interventions: Other: IntelliSpace Precision Medicine Multidisciplinary Team Orchestrator

INTERVENTIONS:
Other: IntelliSpace Precision Medicine Multidisciplinary Team Orchestrator — Digital decision support
  Groups: ISPM -MiProstate

SUMMARY:
This is an observational cohort study with a non-concurrent comparison group evaluating the use of a digital decision support tool (MiProstate/ISPM) at pre-prostatectomy, multidisciplinary conferences.

DETAILED DESCRIPTION:
In the study cohort, all clinically relevant data on patients undergoing radical prostatectomy at Karolinska University Hospital were registered on the platform and subsequently presented using the platform at the conferences in which a detailed treatment plan was devised for each patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients planned for prostatectomy and discussed at pre-operative conference at Karolinska University Hospital

Exclusion Criteria:

-

Sex: Male
Age Groups: Child, Adult, Older Adult
Study Population: Prostate cancer patients at Karolinska University Hospital in the time period Feb 2017- Mar 2019
Sampling Method: Non-Probability Sample
Enrollment: 1329 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Efficiency - time spent in pre-operative conference | Recorded at pre-operative conference held <30 days prior to surgery
  Time spent per patient in pre-operative, multidisciplinary conference, measured by an external observer. After prostate cancer diagnosis, work-up, and the decision to offer the patient surgical treatment with curative intent, a conference is held in which surgical strategies are discussed.
Pre-operative conference quality | Recorded at pre-operative conference held <30 days prior to surgery
  Quality of pre-operative conference as measured by MDT-MODe (MultiDisciplinary Therapy conference - Metric Of Decision Making) score assigned by an external observer. After prostate cancer diagnosis, work-up, and the decision to offer the patient surgical treatment with curative intent, a conference is held in which surgical strategies are discussed.

SECONDARY OUTCOMES:
PSM - positive surgical margin | At surgery. Reported within 30 days after surgery
  Percent of patients with positive surgical margins (an indication of non-radical surgical treatment) as assessed by uro-pathologists
PROM1 - patient-reported outcome measure on urinary function | At 12 months post surgery (11-18 months is tolerated)
  Patient-reported sequelae with respect to urinary function. The Swedish national prostate cancer PROM questionnaire is used. Urinary incontinence is defined as reporting use of one or more protective pads per day.
PROM2 -patient-reported outcome measure on erectile function | At 12 months post surgery (11-18 months is tolerated)
  Patient-reported sequelae with respect to erectile function. The Swedish national prostate cancer PROM questionnaire is used. Erectile dysfunction is defined as IIEF-5 score<12.
Nerve-sparing strategy | Recorded at pre-operative conference (<30 days prior to surgery)
  The nerve-sparing (ns) strategy chosen is reported, specifically percent of patients for which non-ns, uni-lateral or bi-lateral ns procedures are chosen, respectively. Furthermore, the chosen side-specific surgical distance to the prostate is reported as percent intra-fascial ns, inter-fascial ns, semi-ns and non-ns respectively (in increasing order of distance from the prostate capsule).
PLND - pelvic lymph node dissection strategy | Recorded at pre-operative conference (<30 days prior to surgery)
  The frequency of patients for which a decision is made at the pre-operative conference to remove the pelvic lymph nodes (yes/no) is reported

CONTACTS AND LOCATIONS:
Overall Officials: Olof Akre, MD,Professor, Principal Investigator — Karolinska University Hospital, Dept of Pelvic Cancer
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No